CLINICAL TRIAL: NCT06293079
Title: The Effect of Hybrid Telerehabilitation-Based Structured Exercise Programs on Gait, Functional Capacity, EMG Muscle Activation and Fatigue in Patients With Multiple Sclerosis
Brief Title: The Effect of Hybrid Telerehabilitation-Based Structured Exercise Programs in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BiruniUnive; Researcher (Other: Biruni University)
Record Dates: First submitted 2024-02-16; First posted 2024-03-05 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: telerehabilitation; exercise therapy; MS patients
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation Group (Active Comparator): An eight-week rehabilitation program will be implemented synchronously with the physiotherapist two days a week via video conferencing system.
  Interventions: Other: Exercise Program
- Hybrid Telerehabilitation Group (Experimental): The first two weeks of the eight-week program will be applied face to face in the clinic, and the six weeks will be applied synchronously with the physiotherapist via video conferencing system.
  Interventions: Other: Exercise Program
- Clinic Group (Active Comparator): An eight-week rehabilitation program will be implemented face to face in the clinic.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Structured rehabilitation program of the groups; Patient education consists of aerobic and strengthening exercises. An information brochure will be given to patients after the first evaluation about the program to be implemented.

SUMMARY:
The aim of our study is to compare the effects of hybrid telerehabilitation (TR)-based exercise program applied in patients with MS, only TR-based exercise program and only clinical-based exercise program on walking speed, functional capacity, peripheral muscle saturation and fatigue. Forty-five individuals with MS with EDSS scores between 0-4 will be included in the study. The patients will be randomized into three groups: Group A, Group B, and Group C. Group A- Telerehabilitation group will be included in an aerobic and strengthening exercise program over the synchronized videoconference system with the physiotherapist 2 days a week for 8 weeks. Group B- Hybrid Telerehabilitation group will be included in the same exercise program 2 days a week for 2 weeks in the clinic, and will continue remotely over the synchronized videoconference system with the physiotherapist 2 days a week for 6 weeks. In Group C-Clinical Based Rehabilitation group, the same exercise program will be applied in the clinic 2 days a week for 8 weeks. In addition to aerobic and strengthening exercises, traditional breathing exercises and energy conservation techniques will be taught to all three groups within the scope of patient education Demographic and clinical information of all patients to be included in the study will be recorded with a "Case Evaluation Form". The gait speed of the patients will be evaluated with the Timed 25-step walking test, their functional capacity with the 6-minute walking test, their Quadriceps muscle activation will be tested with the EMG muscle activation, the fatigue will be evaluated with the "Modified Fatigue Impact Scale", and the Patient Satisfaction with the "Global Rating Scale". In addition, feasibility evaluation will be made by calculating the attendance rate of the patients to the programs. All data will be evaluated by statistical analysis methods.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic progressive disease that often leads to deterioration of health-related quality of life, including symptoms such as muscle weakness, extreme fatigue, gait disturbances, sensory problems, balance problems, and chronic pain, cognitive and motor impairments. Physiotherapy and rehabilitation programs that include aerobic and progressive resistance exercises in the treatment of functional disorders by controlling the symptoms of the disease increase the quality of life by improving aerobic capacity, but sustainability can be difficult due to difficulties in accessing the clinic. Following exercise programs with telerehabilitation (TR) methods improves cognitive function, mobility, balance, participation, and quality of life by increasing physical activity and reducing fatigue. However, the details of the frequency, duration, and the way the program is delivered are not known, and although the exercise methods applied with TR methods are found to be as effective as the practices performed in the clinic, the remote limited patient-therapist relationship creates potential problems for patients to follow up on the digital platform. The hybrid TR model, in which a certain part of the exercise program is carried out face-to-face, can provide a solution to these problems by increasing patient-therapist communication. To the best of our knowledge, there is no study examining the effectiveness of a rehabilitation program applied with the hybrid TR model for individuals with MS. The aim of our study is to compare the effects of hybrid telerehabilitation (TR)-based exercise program applied in patients with MS, only TR-based exercise program and only clinical-based exercise program on walking speed, functional capacity, peripheral muscle saturation and fatigue. Forty-five individuals with MS with EDSS scores between 0-4 will be included in the study. The patients will be randomized into three groups: Group A, Group B, and Group C. Group A- Telerehabilitation group will be included in an aerobic and strengthening exercise program over the synchronized videoconference system with the physiotherapist 2 days a week for 8 weeks. Group B- Hybrid Telerehabilitation group will be included in the same exercise program 2 days a week for 2 weeks in the clinic, and will continue remotely over the synchronized videoconference system with the physiotherapist 2 days a week for 6 weeks. In Group C-Clinical Based Rehabilitation group, the same exercise program will be applied in the clinic 2 days a week for 8 weeks. In addition to aerobic and strengthening exercises, traditional breathing exercises and energy conservation techniques will be taught to all three groups within the scope of patient education Demographic and clinical information of all patients to be included in the study will be recorded with a "Case Evaluation Form". The gait speed of the patients will be evaluated with the Timed 25-step walking test, their functional capacity with the 6-minute walking test, their Quadriceps muscle activation will be tested with the EMG muscle activation, the fatigue will be evaluated with the "Modified Fatigue Impact Scale", and the Patient Satisfaction with the "Global Rating Scale". In addition, feasibility evaluation will be made by calculating the attendance rate of the patients to the programs. All data will be evaluated by statistical analysis methods. The aim of this study is to investigate the effect of hybrid telerehabilitation program on walking speed, functional capacity, peripheral muscle activation and fatigue in patients with MS.

For these purposes:

* To increase compliance and participation of MS patients in exercises,
* To prevent fatigue by increasing the functional capacity of MS patients who regularly participate in exercise programs,
* To provide a sustainable program for exercise continuity for MS patients who have difficulty reaching the clinic and to examine its effects on fatigue,
* To compare the effects of Telerehabilitation, Hybrid Telerehabilitation and the same exercise programs performed in the clinic on gait speed, functional capacity, peripheral muscle activation and fatigue,
* To examine the statistical differences and relationships between the expected improvements in functional capacity, peripheral muscle activation and fatigue parameters,
* To offer an innovative and effective treatment option to clinicians and experts working in the relevant field with the hybrid telerehabilitation model, which can be an alternative to traditional methods,
* It is aimed to contribute to the literature in this field by transforming the results obtained because of the study into qualified scientific publications.

ELIGIBILITY:
Inclusion Criteria:

* EDSS score of 0 - 4.0
* Having high-speed internet access via smartphone or computer
* Getting at least 24 points from the Mini Mental Test
* Being at Stage 3 or above according to the Functional Ambulation Scale.

Exclusion Criteria:

* Having hearing or vision problems.
* Participating in any exercise program.
* Having other accompanying neurological, cardiovascular or orthopedic disorders
* A history of MS attacks or a change in medication in the last 6 months.
* Being in a physical condition that cannot do the exercises.
* Comorbid conditions that negatively affect oxygen transport (severe anemia, peripheral artery diseases, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Gait Speed | 5 minutes
  The primary evaluation criterion is walking speed. The timed 25-step walking test will be used to evaluate walking speed. In T25FW, which evaluates lower extremity function, patients are asked to walk a distance of 7.62 m as quickly as possible, but without running and safely, and the completion time is recorded in seconds. The average of the two trials is recorded as the T25FW score. T25FW is the best-defined measurement method for measuring gait impairment in individuals with MS and for evaluating the walking speed of patients with gait impairment in the clinical setting
Functional Capacity | 6 minutes
  Functional capacity will be evaluated with a six-minute walk test. The six-minute walk test is a frequently used test that evaluates physical function and walking capacity in patients with MS. According to the principles of the American Thoracic Society, the 6-minute walk test should be performed in the clinic in a 30-meter, flat and hard corridor. The distance walked by the patient is calculated. Patients may stop or slow down if they feel dyspnea. These and similar explanations should be made to the patients. The Borg Dyspnea Scale level, saturation, pulse and blood pressure values should be recorded at the beginning and end of the test.

SECONDARY OUTCOMES:
EMG muscle activation for work and rest average | 5 minutes
  Rectus Femoris and Vastus lateralis muscle activation will be tested with surface EMG device(Myoplus 2 pro)
  During activation and relaxation of muscle; work average time, during rest; rest average time , average release time will be recorded.
EMG muscle activation for peak torque | 5 minutes
  Rectus Femoris and Vastus lateralis muscle activation will be tested with surface EMG device(Myoplus 2 pro)
  During activation and relaxation of muscle; peak torque will be recorded.
Modified Fatigue Impact Scale | 5 minutes
  It is a fatigue scale frequently used in clinical and experimental studies. It evaluates the physical, cognitive and social effects of fatigue. It consists of a total of 21 questions. Each item is given a score between 0 and 4, and a low score indicates a low degree of fatigue. A Turkish validity and reliability study of the this scale has been conducted, and it will be used to determine the fatigue effect in our study

OTHER OUTCOMES:
Global Rating of Change Scale | 1minutes
  Evaluation of Patient Satisfaction: Patient satisfaction will be evaluated with the Global Change Scale. Participants will be asked to express the difference in improvement in their health after treatment compared to before treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Momsen AH, Ortenblad L, Maribo T. Effective rehabilitation interventions and participation among people with multiple sclerosis: An overview of reviews. Ann Phys Rehabil Med. 2022 Jan;65(1):101529. doi: 10.1016/j.rehab.2021.101529. Epub 2022 Jan 25. PMID 33940247
- [Background] Kjolhede T, Vissing K, Langeskov-Christensen D, Stenager E, Petersen T, Dalgas U. Relationship between muscle strength parameters and functional capacity in persons with mild to moderate degree multiple sclerosis. Mult Scler Relat Disord. 2015 Mar;4(2):151-8. doi: 10.1016/j.msard.2015.01.002. Epub 2015 Jan 12. PMID 25787191
- [Background] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Background] Manjaly ZM, Harrison NA, Critchley HD, Do CT, Stefanics G, Wenderoth N, Lutterotti A, Muller A, Stephan KE. Pathophysiological and cognitive mechanisms of fatigue in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2019 Jun;90(6):642-651. doi: 10.1136/jnnp-2018-320050. Epub 2019 Jan 25. PMID 30683707
- [Background] Morris ME, Cantwell C, Vowels L, Dodd K. Changes in gait and fatigue from morning to afternoon in people with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2002 Mar;72(3):361-5. doi: 10.1136/jnnp.72.3.361. PMID 11861697
- [Background] Kos D, Kerckhofs E, Nagels G, D'hooghe MB, Ilsbroukx S. Origin of fatigue in multiple sclerosis: review of the literature. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):91-100. doi: 10.1177/1545968306298934. Epub 2007 Apr 4. PMID 17409388
- [Background] Rottoli M, La Gioia S, Frigeni B, Barcella V. Pathophysiology, assessment and management of multiple sclerosis fatigue: an update. Expert Rev Neurother. 2017 Apr;17(4):373-379. doi: 10.1080/14737175.2017.1247695. Epub 2016 Oct 21. PMID 27728987
- [Result] Tollar J, Nagy F, Toth BE, Torok K, Szita K, Csutoras B, Moizs M, Hortobagyi T. Exercise Effects on Multiple Sclerosis Quality of Life and Clinical-Motor Symptoms. Med Sci Sports Exerc. 2020 May;52(5):1007-1014. doi: 10.1249/MSS.0000000000002228. PMID 31876670